CLINICAL TRIAL: NCT05709847
Title: The Effects of CGA-rich Coffee on Cognitive Function in Type 2 Diabetes: A Parallel Groups Randomised Controlled Trial
Brief Title: The Effects of Specialty Coffee on Cognitive Function in People With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Daniel Lamport, Associate Professor Daniel Lamport, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UReading Coffee Diabetes Study
Record Dates: First submitted 2022-11-11; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Coffee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional coffee (Active Comparator): Participants will be provided with a conventional, low CGA coffee to brew and consume which contains less CGA than the experimental arm.
  Interventions: Other: Coffee
- CGA-rich coffee (Speciality coffee) (Experimental): Participants will be provided with a single origin, CGA-rich specialty coffee as graded by the Specialty Coffee Association of America's Q-grading system to brew and consume
  Interventions: Other: Coffee

INTERVENTIONS:
Other: Coffee — 24 ounces of coffee will be consumed daily

SUMMARY:
Coffee has been found to have beneficial effects on cognitive function and blood sugar control. Benefits include reduced risk of cognitive decline and improved performance on cognitive tests, as well as reduced risk of diabetes and improved blood sugar control in people with diabetes, a population that is at a higher risk of cognitive decline. These effects have been observed for both caffeinated and decaffeinated coffee, and have been associated with the polyphenol chlorogenic acid (CGA). This polyphenol has been found to be more bioavailable in certain coffees, known as "speciality coffee" as defined by the Specialty Coffee Association of America, depending on agriculture, roasting, and brewing method.

This current project will bring together these previous findings to explore the effects of specialty coffee on cognitive function and glycaemic control in people with type 2 diabetes through a randomized control trial with two groups: a high CGA specialty coffee group and a conventional coffee control group. Participants will be quasi-randomly assigned to one of these two groups following the completion of a 4-week run-in period during which participants will consume conventional coffee only. The length of the experimental arms is 8 weeks, therefore the total length of the study is 12 weeks. At the beginning and the end of each experimental arm participants will undertake a cognitive assessment online using the Gorilla platform, and a series of questionnaires relating to health and mood measures (details in procedure). Cognitive function will also be assessed at the beginning of the 4-week run-in period.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-70 years
* Formal diagnosis of Type 2 Diabetes for 3 years or more
* Current coffee drinkers, 4 or fewer cups daily (a cup is 8 oz)

Exclusion Criteria:

* Insulin-dependent
* Consuming on average more than 4 cups of coffee daily
* Regularly consuming specialty coffee (participants will be provided with a list of these coffees)

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Verbal memory | 8 weeks
  Assessed at the end of 8-week intervention arm using a modified version of the Rey Auditory Verbal Learning Test
Verbal memory | 0 weeks
  Assessed at the beginning of the 8-week intervention arm using a modified version of the Rey Auditory Verbal Learning Test
Verbal memory | -4 weeks
  Assessed at the beginning of the 4-week run-in period using a modified version of the Rey Auditory Verbal Learning Test

SECONDARY OUTCOMES:
Haemoglobin A1C | 8 weeks
  Self-reported by the participant at the end of the 8-week intervention arm
Haemoglobin A1C | 0 weeks
  Self-reported by the participant at the beginning of the 8-week intervention arm
Haemoglobin A1C | -4 weeks
  Self-reported by the participant at the beginning of the 4-week run-in period
Lipid panel (total cholesterol, HDL, LDL, triglycerides) | 8 weeks
  Self-reported by the participant at the end of the 8-week intervention arm
Lipid panel (total cholesterol, HDL, LDL, triglycerides) | 0 weeks
  Self-reported by the participant at the beginning of the 8-week intervention arm
Lipid panel (total cholesterol, HDL, LDL, triglycerides) | -4 weeks
  Self-reported by the participant at the beginning of the 4-week run-in period
Depression symptoms | 8 weeks
  Assessed at the end of the 8-week intervention arm with the PHQ-9
Depression symptoms | 0 weeks
  Assessed at the beginning of the 8-week intervention arm with the PHQ-9
Depression symptoms | -4 weeks
  Assessed at the beginning of the 4-week run-in period with the PHQ-9
Anxiety symptoms | 8 weeks
  Assessed at the end of the 8-week intervention arm with the GAD-7
Anxiety symptoms | 0 weeks
  Assessed at the beginning of the 8-week intervention arm with the GAD-7
Anxiety symptoms | -4 weeks
  Assessed at the beginning of the 4-week run-in period with the GAD-7
Executive Function | 8 weeks
  Assessed at the end of the 8-week intervention arm with a computerised version of the Corsi Block Tapping Test
Executive Function | 0 weeks
  Assessed at the beginning of the 8-week intervention arm with a computerised version of the Corsi Block Tapping Test
Executive Function | -4 weeks
  Assessed at the beginning of the 4-week run-in with a computerised version of the Corsi Block Tapping Test
Working memory | 0 weeks
  Assessed at the beginning of the 8-week intervention arm with a computerised version of digit span
Working memory | -4 weeks
  Assessed at the beginning of the 4-week run-in with a computerised version of digit span
Processing Speed | 8 weeks
  Assessed at the end of the 8-week intervention arm with a computerised version of the Digit Symbol Substitution Test
Processing Speed | 0 weeks
  Assessed at the beginning of the 8-week intervention arm with a computerised version of the Digit Symbol Substitution Test
Processing Speed | -4 weeks
  Assessed at the beginning of 4-week run-in with a computerised version of the Digit Symbol Substitution Test

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lamport, PhD, Principal Investigator — University of Reading
Locations (1):
- Kaiser Permanente, Berkeley, California, United States